CLINICAL TRIAL: NCT03385148
Title: Diagnostic Performance and Evaluation Efficacy of a Novel PTK7 PET Radiotracer 68Ga-SGC8
Brief Title: The Clinical Application of 68Ga Labeled ssDNA Aptamer Sgc8 in Healthy Volunteers and Colorectal Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20162077-2
Record Dates: First submitted 2017-12-19; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- colorectal patients (Experimental): the colorectal patients undergo 68Ga-Sgc8 PET/CT
  Interventions: Drug: 68Ga-Sgc8

INTERVENTIONS:
Drug: 68Ga-Sgc8 — underwent a standard routine 18F-FDG PET/CT first, and then injected 10~20 MBq 68Ga-Sgc8
  Other Names: PET/CT

SUMMARY:
The protein tyrosine kinase-7 (PTK7) is overexpressed in various types of human cancers. As a specific imaging agent of PTK7, 68Ga-Sgc8 was investigated in this study to assess its safety, biodistribution and dosimetric properties in healthy volunteers, and to preliminarily evaluate its application in colorectal patients.

DETAILED DESCRIPTION:
The protein tyrosine kinase-7 (PTK7), also known as colon carcinoma kinase-4 (CCK4), is a member of the receptor tyrosine kinase superfamily, which is evolutionarily conserved and contains seven immunoglobulin domains, a transmembrane domain, and a catalytically inactive kinase domain. PTK7 controls tissue morphogenesis and patterning by affecting cell polarity, migration as well as tissue regeneration and wound healing. It's reported that PTK7 plays an important role in the motility and invasivity of cancer cells and is overexpresses in many different types of human cancers, including colon, lung, gastric, breast cancer etc, making it a potentially attractive target for quantitative imaging and therapy.

Sgc8, a 41 oligonucleotides single-stranded DNA aptamer, which was selected by cell based systematic evolution of ligands by exponential enrichment (SELEX), has been identified as a specific ligand of PTK7. In this study, Sgc8 was linked to a bi-functional group NOTA for 68Ga chelation. The previous studies showed that the Sgc8 derivatives have a high accumulation in PTK7 positive tumors, suggesting the feasibility of 68Ga-Sgc8 for clinical translation for cancer detection.

Colorectal cancer (CRC) represents the third common type of cancer and the fourth leading cause of death in the worldwide, and has one of the highest rates of synchronous or metachronous malignancy among all cancers. According to the Colon Cancer NCCN Guidelines (version 3.2014), 50-60% CRC patients are with metastases, and 80-90% of these metastatic patients may have unresectable liver metastasis. Therefore, early detection of the lesions is of utmost importance with respect to administration of early treatment and improved survival. It's reported that PTK7 is overexpressed in CRC, and the expression was correlated with tumor differentiation, lymph node metastasis, distant metastasis and TNM stage of CRC patients, suggesting that PTK7 may be a desirable target to predict the occurrence and prognosis of colorectal tumor.

In this study, investigators will first measur the dosimetry of 68Ga-Sgc8 in healthy volunteers, and then evaluate the tracer in colorectal patients, to assess its diagnostic value.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent
* Males and females, ≥18 years old；
* Newly diagnosed colorectal patients and lymph node metastasis is not clear. The tumor will be surgically removed and histological diagnosis will be available.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential；
* Known severe allergy or hypersensitivity to IV radiographic contrast；
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
diagnosis effecacy | 2 years
  Assess advantage or concordance of 68Ga-Sgc8 PET results with 18F-FDG PET imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, Dr., Study Chair — Xijing Hospital
Locations (2):
- China (2):
  - Xijing Hospital Nuclear Medicine Department, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No